CLINICAL TRIAL: NCT05457556
Title: A Multi-Center, Phase 3, Randomized Trial of Matched Unrelated Donor (MUD) Versus HLA-Haploidentical Related (Haplo) Myeloablative Hematopoietic Cell Transplantation for Children, Adolescents, and Young Adults (AYA) With Acute Leukemia or Myelodysplastic Syndrome (MDS)
Brief Title: Mismatched Related Donor Versus Matched Unrelated Donor Stem Cell Transplantation for Children, Adolescents, and Young Adults With Acute Leukemia or Myelodysplastic Syndrome
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASCT2031; NCI-2022-07080 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ASCT2031 (Other: Children's Oncology Group); ASCT2031 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2022-07-11; First posted 2022-07-14 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-05

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Mixed Phenotype Acute Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute; Myelodysplastic Syndromes | interventions — Specimen Handling; Busulfan; Cyclophosphamide; fludarabine; Stem Cell Transplantation; Antilymphocyte Serum; thymoglobulin; Spinal Puncture; Melphalan; Methotrexate; merphos; Mycophenolic Acid; Bone Marrow Purging; Rituximab; CT-P10; Tacrolimus; Thiotepa; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm A (halploHCT) (Experimental): Patients receive a myeloablative conditioning regimen with PTCy or alpha beta T cell depletion at the discretion of the treating provider. Patients then undergo haploHCT on day 0. Patients undergoing myeloablative conditioning regimen with PTCy also receive GVHD prophylaxis on days 3-5. Patients undergo lumbar puncture, bone marrow aspiration, and ECHO or MUGA during screening. Patients also undergo collection of blood throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Drug: Busulfan; Drug: Cyclophosphamide; Procedure: Echocardiography Test; Drug: Fludarabine; Procedure: Haploidentical Hematopoietic Cell Transplantation; Biological: Lapine T-Lymphocyte Immune Globulin; Procedure: Lumbar Puncture; Drug: Melphalan; Procedure: Multigated Acquisition Scan; Drug: Mycophenolate Mofetil; Procedure: Myeloablative Conditioning; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Biological: Rituximab; Procedure: T-Cell Depletion Therapy; Drug: Tacrolimus; Drug: Thiotepa; Radiation: Total-Body Irradiation
- Arm B (MUD-HCT) (Experimental): Patients receive a TBI-based or chemotherapy-based myeloablative conditioning regimen between days -9 and -2, followed by MUD-HCT on day 0. Patients then receive GVHD prophylaxis regimen on days 1-11. Patients undergo lumbar puncture, bone marrow aspiration, and ECHO or MUGA during screening. Patients also undergo collection of blood throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Drug: Busulfan; Drug: Cyclophosphamide; Procedure: Echocardiography Test; Drug: Fludarabine; Biological: Lapine T-Lymphocyte Immune Globulin; Procedure: Lumbar Puncture; Procedure: Matched Unrelated Donor Hematopoietic Cell Transplantation; Drug: Methotrexate; Procedure: Multigated Acquisition Scan; Procedure: Myeloablative Conditioning; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Tacrolimus; Drug: Thiotepa; Radiation: Total-Body Irradiation
- Arm C (haploHCT) (Experimental): Patients who only have a haplo donor receive a myeloablative conditioning regimen with PTCy or alpha beta T cell depletion at the discretion of the treating provider. Patients then undergo haploHCT on day 0. Patients undergoing myeloablative conditioning regimen with PTCy also receive GVHD prophylaxis on days 3-5. Patients undergo lumbar puncture, bone marrow aspiration, and ECHO or MUGA during screening. Patients also undergo collection of blood throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Drug: Busulfan; Drug: Cyclophosphamide; Procedure: Echocardiography Test; Drug: Fludarabine; Procedure: Haploidentical Hematopoietic Cell Transplantation; Biological: Lapine T-Lymphocyte Immune Globulin; Procedure: Lumbar Puncture; Drug: Melphalan; Procedure: Multigated Acquisition Scan; Drug: Mycophenolate Mofetil; Procedure: Myeloablative Conditioning; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Biological: Rituximab; Procedure: T-Cell Depletion Therapy; Drug: Tacrolimus; Drug: Thiotepa; Radiation: Total-Body Irradiation

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration
Drug: Busulfan — Given intravenously (IV)
  Other Names: 1, 4-Bis[methanesulfonoxy]butane; BUS; Busilvex; Bussulfam; Busulfanum; Busulfex; Busulphan; CB 2041; CB-2041; Glyzophrol; GT 41; GT-41; Joacamine; Methanesulfonic Acid Tetramethylene Ester; Methanesulfonic acid, tetramethylene ester; Mielucin; Misulban; Misulfan; Mitosan; Myeleukon; Myeloleukon; Myelosan; Mylecytan; Myleran; Sulfabutin; Tetramethylene Bis(methanesulfonate); Tetramethylene bis[methanesulfonate]; WR-19508
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Asta B 518; B 518; B-518; B518; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR 138719; WR- 138719; WR-138719; WR138719
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Procedure: Haploidentical Hematopoietic Cell Transplantation — Undergo haploHCT
  Other Names: Haploidentical Stem Cell Transplantation; HLA-Haploidentical Hematopoietic Cell Transplantation; Stem Cell Transplantation, Haploidentical
  Arms: Arm A (halploHCT); Arm C (haploHCT)
Biological: Lapine T-Lymphocyte Immune Globulin — Given IV
  Other Names: Anti-Thymocyte Globulin Rabbit; Antithymocyte Globulin Rabbit; Antithymocyte globulin rabbit ATG; Grafalon; Imtix; Rabbit Anti-Human Thymocyte Globulin (RATG); Rabbit Anti-Thymocyte Globulin; Rabbit Antithymocyte Globulin; Rabbit ATG; Thymoglobulin
Procedure: Lumbar Puncture — Undergo lumbar puncture
  Other Names: LP; Spinal Tap
Procedure: Matched Unrelated Donor Hematopoietic Cell Transplantation — Undergo MUD-HCT
  Other Names: MUD-HCT
  Arms: Arm B (MUD-HCT)
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalan for Injection-Hepatic Delivery System; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
  Arms: Arm A (halploHCT); Arm C (haploHCT)
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Jylamvo; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
  Arms: Arm B (MUD-HCT)
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Mycophenolate Mofetil — Given IV
  Other Names: CellCept; MMF
  Arms: Arm A (halploHCT); Arm C (haploHCT)
Procedure: Myeloablative Conditioning — Receive myeloablative conditioning regimen
  Other Names: Myeloablation; Myeloablative; Myeloablative Cytoreduction
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Biological: Rituximab — Given IV
  Other Names: ABP 798; ABP-798; ABP798; BI 695500; BI-695500; BI695500; Blitzima; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT P10; CT-P10; CTP10; GP 2013; GP-2013; GP2013; IDEC 102; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; IDEC102; Ikgdar; Mabtas; MabThera; Monoclonal Antibody IDEC-C2B8; PF 05280586; PF-05280586; PF05280586; Riabni; Ritemvia; Rituxan; Rituximab ABBS; Rituximab ARRX; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar GP2013; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; Rituximab PVVR; Rituximab-abbs; Rituximab-arrx; Rituximab-blit; Rituximab-pvvr; Rituximab-rite; Rituximab-rixa; Rituximab-rixi; Rixathon; Riximyo; RTXM 83; RTXM-83; RTXM83; Ruxience; Truxima
  Arms: Arm A (halploHCT); Arm C (haploHCT)
Procedure: T-Cell Depletion Therapy — Undergo haploHCT with alpha beta T cell depletion
  Other Names: T-Cell Depletion; T-Lymphocyte Depletion Therapy
  Arms: Arm A (halploHCT); Arm C (haploHCT)
Drug: Tacrolimus — Given IV
  Other Names: FK 506; FK-506; FK506; Fujimycin; Hecoria; Prograf; Protopic; Tacforius
Drug: Thiotepa — Given IV
  Other Names: 1,1',1''-Phosphinothioylidynetrisaziridine; Girostan; N,N', N''-Triethylenethiophosphoramide; Oncotiotepa; SH 105; SH-105; SH105; STEPA; Tepadina; Tepylute; TESPA; Tespamin; Tespamine; Thio-Tepa; Thiofosfamide; Thiofozil; Thiophosphamide; Thiophosphoamide; Thiophosphoramide; Thiotef; Tifosyl; TIO TEF; Tio-tef; Triethylene Thiophosphoramide; Triethylenethiophosphoramide; Tris(1-aziridinyl)phosphine sulfide; TSPA; WR 45312
Radiation: Total-Body Irradiation — Undergo TBI
  Other Names: SCT_TBI; TBI; Total Body Irradiation; Whole Body; Whole Body Irradiation; Whole-Body Irradiation

SUMMARY:
This phase III trial compares hematopoietic (stem) cell transplantation (HCT) using mismatched related donors (haploidentical [haplo]) versus matched unrelated donors (MUD) in treating children, adolescents, and young adults with acute leukemia or myelodysplastic syndrome (MDS). HCT is considered standard of care treatment for patients with high-risk acute leukemia and MDS. In HCT, patients are given very high doses of chemotherapy and/or radiation therapy, which is intended to kill cancer cells that may be resistant to more standard doses of chemotherapy; unfortunately, this also destroys the normal cells in the bone marrow, including stem cells. After the treatment, patients must have a healthy supply of stem cells reintroduced or transplanted. The transplanted cells then reestablish the blood cell production process in the bone marrow. The healthy stem cells may come from the blood or bone marrow of a related or unrelated donor. If patients do not have a matched related donor, doctors do not know what the next best donor choice is. This trial may help researchers understand whether a haplo related donor or a MUD HCT for children with acute leukemia or MDS is better or if there is no difference at all.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the 1-year cumulative incidence of severe Graft Versus Host Disease (GVHD) (from day of HCT) defined as grade III-IV acute GVHD (aGVHD) and/or chronic GVHD (cGVHD) that requires systemic immunosuppression and to compare the disease free survival (DFS) (from time of randomization) in children and young adults (AYA) with acute myeloid leukemia (AML), acute lymphoid leukemia (ALL), mixed phenotype acute leukemia (MPAL), and myelodysplastic syndrome (MDS) who are randomly assigned to haploHCT or to an 8/8 adult MUD-HCT.

SECONDARY OBJECTIVES:

I. To compare overall survival (OS) between children and AYA with AML/ALL/MPAL/MDS randomly assigned to haploHCT and MUD HCT.

II. To compare differences in health-related quality of life (HRQOL) between haploHCT and MUD HCT from baseline (pre-transplant), at 6 months, 1 year and 2 years post-transplant.

EXPLORATORY OBJECTIVES:

I. To compare the median time to engraftment and cumulative incidences of neutrophil engraftment at 30 and 100 days post transplant and platelet engraftment at 60 and 100 days post transplant, primary graft failure by 60 days, secondary graft failure at 1 year post transplant, Grade II-IV and III-IV acute graft versus host disease (aGVHD) requiring systemic immunosuppression at 100 days and 6 months, and cumulative incidences of transplant-related mortality (TRM), relapse, and moderate and severe chronic graft versus host disease (cGVHD) at 6 months, 1 and 2 years after haploHCT and MUD HCT.

II. To estimate 1 year, 18-month and 2-year cumulative incidence of graft-versus-host disease (GVHD)-free relapse-free survival (GRFS) with events defined as occurrence of any of the following from Day 0 of HCT: Grade III-IV acute GVHD, chronic GVHD requiring systemic immunosuppressive treatment, disease relapse or progression, and death from any cause.

IIa. To compare "chronic GVHD" (GRFS) after haploHCT and MUD HCT using landmark definitions.

IIb. To compare "current" GRFS is defined as the time to onset of any of the following events from Day 0 of HCT: Grade III-IV acute GVHD, chronic GVHD that is STILL requiring systemic immunosuppressive treatment, disease relapse or progression, death from any cause at 18 months and 2 years.

III. To evaluate the influence of key clinical variables: age (<13 years and 13-21.99 years), disease (ALL/MPAL versus [vs.] AML/MDS), haploHCT approach (TCR alpha beta + T cell depletion vs. post-transplant cyclophosphamide [PTCy]); donor age (by ten-year increments), donor sex (maternal vs. paternal for parental donation), pre-HCT minimal residual disease status (MRD + vs MRD -); pediatric disease risk index (low, intermediate, and high, impact on OS and DFS only), conditioning regimen (chemotherapy based versus total-body irradiation [TBI] based), immunosuppressive regimen (anti-thymocyte globulin [ATG] exposure according to the weight and absolute lymphocyte count [ALC] dependent dosing approach vs no ATG exposure) time to transplant (interval between diagnosis/relapse and date of stem cell infusion) graft cell dose, use of relapse prevention therapy (yes or no) and weight on engraftment, OS, DFS, GRFS, relapse, transplant related mortality (TRM), aGvHD and cGvHD at 1 and 2 years after haplo and MUD HCT by performing stratified and multivariate analyses.

IV. To compare other important transplant related outcomes after haplo and MUD HCT, such as:

IVa. Incidence of any significant fungal infections (defined as proven or probable fungal infection) through 1 year post HCT; IVb. Incidence of viremia with or without end organ disease (i.e. cytomegalovirus [CMV], adenovirus, Epstein-Barr virus [EBV], human herpesvirus 6 [HHV-6], BK) requiring hospitalization and/or systemic antiviral therapy and/or cell therapy through 1 year post HCT; IVc. Incidence of sinusoidal obstruction syndrome (SOS) through 100 days post HCT; IVd. As defined by the Cairo criteria; IVe. To compare the incidence and outcome of SOS when different criteria are used (European Bone Marrow Transplant [EBMT], Cairo, Baltimore, and modified Seattle criteria); IVf. Incidence of transplant-associated thrombotic microangiopathy (TA-TMA) through 100 days post HCT.

V. To compare immune recovery after haplo PTCy, haplo alpha-beta T cell depletion, and MUD HCT via:

Va. Pace of reconstitution of T, B, and natural killer (NK) cells and immunoglobulins at 30 days, 60 days, 100 days, 180 days and 365 days after HCT; Vb. Response to vaccinations as determined by vaccination-specific antibody titers at 12-18 months post hematopoietic stem cell transplant (HSCT); Vc. Biobanking blood or marrow to analyze the impact of graft composition on GvHD, relapse and viremia; Vd. Biobanking whole blood and serum to compare immune recovery using extended immune phenotyping and immune functional assessments.

VI. Biobanking whole blood or serum to measure rabbit antithymocyte globulin (rATG) exposure when dosed according to weight and absolute lymphocyte count (ALC) using established pharmacokinetic and pharmacodynamics assays (after last infusion, Day -4, Day 0, Day +7).

VII. To compare resource utilization after haplo and MUD HCT. VIIa. Length of HCT hospital stay from Day 0 and readmissions within the first 100 days (number of readmissions, duration, and reason).

VIIb. Inpatient costs within the first 100 days and at 2 years post HCT. VIII. To describe and compare outcomes (neutrophil and platelet engraftment, graft failure, OS, DFS, GRFS, NRM, relapse, GvHD and health-related quality of life [HRQOL] post HCT) by recipient race/ethnicity, annual household income, primary spoken language and conserved transcriptional response to adversity (CTRA).

IX. To describe HRQoL outcomes in racial/ethnic minorities and compare HRQoL outcomes between White patients receiving haploHCT and racial/ethnic minority patients receiving haploHCT.

X. To assess the feasibility of incorporating total body irradiation (TBI) delivered with volumetric modulated arc therapy (VMAT) or tomotherapy into a multi-institutional study, to describe the toxicities and oncologic outcomes (relapse, DFS, OS, and TRM) of the subgroup of patients treated with this approach, and to compare these outcomes to those of patients treated with conventional TBI.

OUTLINE: Patients who have both a MUD and haplo donor are randomized to Arm A or Arm B. Patients who only have a haplo donor are nonrandomly assigned to Arm C.

ARM A: Patients receive a haplo HCT following a TBI- based or chemotherapy-based myeloablative conditioning regimen with PTCy or alpha beta T cell depletion (center's choice). When PTCy is used, it Is administered on days 3 and 4 after HCT and additional immunsouppression is started on day 5 after SCT.

ARM B: Patients receive a MUD HCT following a TBI-based or chemotherapy-based myeloablative conditioning regimen between days -9 and -2 Patients then receive GVHD prophylaxis on days 1-11.

ARM C: Patients receive a haploHCT following a TBI-based or chemotherapy-based myeloablative conditioning regimen with PTCy or alpha beta T cell depletion (center's choice). When PTCy is used, it Is administered on days 3 and 4 after HCT and additional immunsouppression is started on day 5 after SCT.

Patients in all arms undergo standard HCT screening prior to transplant including disease evaluation (lumbar puncture, bone marrow aspiration), and organ function evaluation including but not limited to echocardiogram (ECHO) or multigated acquisition scan (MUGA), PFTS, and bloodwork.Patients also undergo collection of blood throughout the trial.

After completion of study treatment, patients are followed periodically for up to 5 years from HCT.

ELIGIBILITY:
Inclusion Criteria:

* PATIENT INCLUSION CRITERIA FOR ENROLLMENT:
* 6 months to < 22 years at enrollment
* Diagnosed with ALL, AML, or MDS or mixed phenotype acute leukemia (MPAL) for which an allogeneic hematopoietic stem cell transplant is indicated. Complete Remission (CR) status will not be confirmed at the time of enrollment. CR as defined in these sections is required to proceed with the actual HCT treatment plan
* Has not received a prior allogeneic hematopoietic stem cell transplant
* Does not have a suitable human leukocyte antigen (HLA)-matched sibling donor available for stem cell donation
* Has an eligible haploidentical related family donor based on at least intermediate resolution HLA typing

  * Patients who also have an eligible 8/8 MUD adult donor based on confirmatory high resolution HLA typing are eligible for randomization to Arm A or Arm B.
  * Patients who do not have an eligible MUD donor are eligible for enrollment to Arm C
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met
* Co-Enrollment on other trials

  * Patients will not be excluded from enrollment on this study if already enrolled on other protocols for treatment of high risk and/or relapsed ALL, AML, MPAL and MDS. This is including, but not limited to, COG AAML1831, COG AALL1821, the EndRAD Trial, as well as local institutional trials. We will collect information on all co-enrollments
  * Patients will not be excluded from enrollment on this study if receiving immunotherapy prior to transplant as a way to achieve remission and bridge to transplant. This includes chimeric antigen receptor (CAR) T cell therapy and other immunotherapies
* PATIENT INCLUSION CRITERIA TO PROCEED TO HCT:
* Karnofsky Index or Lansky Play-Performance Scale >= 60 on pre-transplant evaluation. Karnofsky scores must be used for patients >= 16 years of age and Lansky scores for patients =< 16 years of age (within 4 weeks of starting therapy)
* A serum creatinine based on age/gender as follows:

  6 months to < 1 year: 0.5 mg/dL (Male); 0.5 mg/dL (Female)
  1. to < 2 years: 0.6 mg/dL (Male); 0.6 mg/dL (Female)
  2. to < 6 years: 0.8 mg/dL (Male); 0.8 mg/dL (Female)

  6 to < 10 years: 1 mg/dL (Male); 1 mg/dL (Female) 10 to < 13 years: 1.2 mg/dL (Male); 1.2 mg/dL (Female) 13 to < 16 years: 1.5 mg/dL (Male); 1.4 mg/dL (Female) >= 16 years: 1.7 mg/dL (Male); 1.4 mg/dL (Female)
  * OR
* A 24 hour urine Creatinine clearance >= 60 mL/min/1.73 m^2

  * OR
* A glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2. GFR must be performed using direct measurement with a nuclear blood sampling method OR direct small molecule clearance method (iothalamate or other molecule per institutional standard)

  * Note: Estimated GFR (eGFR) from serum creatinine, cystatin C or other estimates are not acceptable for determining eligibility
* Serum glutamic-oxaloacetic transaminase (SGOT) aspartate aminotransferase [AST] or serum glutamate pyruvate transaminase (SGPT) aminotransferase [ALT] < 5 x upper limit of normal (ULN) for age
* Total bilirubin < 2.5 mg/dL, unless attributable to Gilbert's Syndrome
* Shortening fraction of >= 27% by echocardiogram or radionuclide scan (MUGA)

  * OR
* Ejection fraction of >= 50% by echocardiogram or radionuclide scan (MUGA), choice of test according to local standard of care
* Forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), and corrected carbon monoxide diffusing capability (DLCO) must all be >= 50% of predicted by pulmonary function tests (PFTs).

  * For children who are unable to perform for PFTs (e.g., due to age or developmental delay), the criteria are: no evidence of dyspnea at rest, oxygen (O2) saturation (Sat) > 92% on room air by pulse oximetry, not on supplemental O2 at rest, and not on supplemental O2 at rest
* MPAL in first complete remission (CR1) for whom transplant is indicated. Examples include those patients who are poorly responsive to ALL therapy (end of induction failure( IF-MPAL) to ALL induction (see IF-MPAL note below), end of induction MRD ≥ 5% or end-of-consolidation MRD > 0.01%), as well as patients treated with AML therapy
* IF-MPAL: additional criterion for Induction failure for MPAL ONLY as per ALL1732:

  * An increasing number of circulating leukemia cells on 3 or more consecutive CBCs obtained at daily or longer intervals following day 8 of Induction therapy and prior to day 29 with confirmation by flow cytometry OR development of new sites of extramedullary disease, or other laboratory or clinical evidence of refractory disease or progression prior to the end of Induction evaluation (note that residual testicular disease at the end of Induction is an exception)
* MPAL in > second complete remission (CR2)
* ALL high-risk in CR1 for whom transplant is indicated. Examples include: induction failure, treatment failure as per minimal residual disease by flow cytometry > 0.01% after consolidation and not eligible for AALL1721 or AALL1721 not available/unwilling to enroll, hypodiploidy (< 44 chromosomes) with MRD+ > 0.01% after induction, persistent or recurrent cytogenetic or molecular evidence of disease during therapy requiring additional therapy after induction to achieve remission (e.g. persistent molecular BCR-ABL positivity), T cell ALL with persistent MRD > 0.01% after consolidation.
* ALL in CR2 for whom transplant is indicated. Examples include: B-cell: early (=< 36 months from initiation of therapy) bone marrow (BM) relapse, late BM relapse (>= 36 months) with MRD >= 0.1% by flow cytometry after first re-induction therapy; T or B-cell: early (< 18 months) isolated extramedullary (IEM), late (>= 18 months) IEM, end-Block 1 MRD >= 0.1%; T-cell or Philadelphia chromosome positive (Ph+): BM relapse at any time
* ALL in >= third complete remission (CR3)
* Patients treated with chimeric antigen receptor T-cells (CART) cells for whom transplant is indicated. Examples include: transplant for consolidation of CART, loss of CART persistence and/or B cell aplasia < 6 months from infusion or have other evidence (e.g., MRD+) that transplant is indicated to prevent relapse
* AML in CR1 for whom transplant is indicated. Examples include those deemed high risk for relapse as described in AAML1831:

  * FLT3/ITD+ with allelic ratio > 0.1 without bZIP CEBPA, NPM1
  * FLT3/ITD+ with allelic ratio > 0.1 with concurrent bZIP CEBPA or NPM1 and with evidence of residual AML (MRD >= 0.05%) at end of Induction
  * Presence of RAM phenotype or unfavorable prognostic markers (other than FLT3/ITD) per cytogenetics, fluorescence in situ hybridization (FISH), next generation sequencing (NGS) results, regardless of favorable genetic markers, MRD status or FLT3/ITD mutation status
  * AML without favorable or unfavorable cytogenetic or molecular features but with evidence of residual AML (MRD >= 0.05%) at end of Induction
  * Presence of a non-ITD FLT3 activating mutation and positive MRD (>= 0.05%) at end of Induction 1 regardless of presence of favorable genetic markers.
* AML in >= CR2
* MDS with < 5% blasts by morphology and flow cytometry (if available) on the pre-transplant bone marrow evaluation
* Complete remission (CR) is defined as < 5% blasts by morphology and flow cytometry (if available) on the pre-transplant bone marrow evaluation with minimum sustained absolute neutrophil count (ANC) of 300 cells/microliter for 1 week or ANC > 500 cells/microliter. We will be collecting data from all approaches to MRD evaluation performed including NGS and polymerase chain reaction (PCR). It is strongly recommended that MPAL be evaluated using multidimensional flow cytometry and/or (KMT2Ar) qt PCR. It is strongly recommended that MPAL be evaluated using multidimensional flow cytometry and/or (KMT2Ar) qt PCR
* DONOR ELIGIBILITY CRITERIA:
* Matched Unrelated Donors:

Unrelated donor candidates must be matched at high resolution at a minimum of 8/8 alleles (HLA-A, -B, -C, -DRB1). One-antigen HLA mismatches are not permitted. HLA matching of additional alleles is recommended according to National Marrow Donor Program (NMDP) guidelines, but will be at the discretion of local centers

* Haploidentical Matched Family Members:

  * Minimum match level full haploidentical (at least 5/10; HLA-A, -B, -C, -DRB1, -DQB1 alleles). The following issues (in no particular order) should be considered in choosing a haploidentical donor:

    * Absent or low patient donor-specific antibodies (DSA)

      * Mean fluorescence intensity (MFI) of any anti-donor HLA antibody by solid phase immunoassay should be < 2000. Donors with higher levels are not eligible.

        * If a screening assay against pooled HLA antigens is used, positive results must be followed with specificity testing using a single antigen assay. The MFI must be < 2000 unless the laboratory has validated higher threshold values for reactivity for HLA antigens (such as HLA-C, -DQ, and -DP), that may be enhanced in concentration on the single antigen assays. Donor anti- recipient antibodies are of unknown clinical significance and do not need to be sent or reported.
        * Consult with Study Chair for the clinical significance of any recipient anti-donor HLA antibody.
        * If centers are unable to perform this type of testing, please contact the Study Chair to make arrangements for testing.
    * If killer immunoglobulin testing (KIR) is performed: KIR status by mismatch, KIR-B, or KIR content criteria can be used according to institutional guidelines.
    * ABO compatibility (in order of priority):

      * Compatible or minor ABO incompatibility
      * Major ABO incompatibility
    * CMV serostatus:

      * For a CMV seronegative recipient: the priority is to use a CMV seronegative donor when feasible
      * For a CMV seropositive recipient: the priority is to use a CMV seropositive donor when feasible
    * Age: younger donors including siblings/half-siblings, and second degree relatives (aunts, uncles, cousins) are recommended, even if < 18 years
* Size and vascular access appropriate by center standard for peripheral blood stem cell (PBSC) collection if needed
* Haploidentical matched family members: screened by center health screens and found to be eligible
* Unrelated donors: meet eligibility criteria as defined by the NMDP or other unrelated donor registries. If the donor does not meet the registry eligibility criteria but an acceptable eligibility waiver is completed and signed per registry guidelines, the donor will be considered eligible for this study
* Human immunodeficiency virus (HIV) negative
* Not pregnant
* MUD donors and post-transplant cyclophosphamide haplo donors should be asked to provide BM. If donors refuse and other donors are not available, PBSC is allowed. TCR-alpha beta/CD19 depleted haplo donors must agree to donate PBSC
* Must give informed consent:

  * Haploidentical matched family members: Institution standard of care donor consent and Protocol-specific Donor Consent for Optional Studies
  * Unrelated donors: standard NMDP Unrelated Donor Consent

Exclusion Criteria:

* PATIENT EXCLUSION CRITERIA FOR ENROLLMENT:
* Patients with genetic disorders (generally marrow failure syndromes) prone to secondary AML/ALL/MPAL with known poor outcomes because of sensitivity to alkylator therapy and/or TBI are not eligible (Fanconi Anemia, Kostmann Syndrome, Dyskeratosis Congenita, etc). Patients with Downs syndrome because of increased toxicity with intensive conditioning regimens.
* Patients with any obvious contraindication to myeloablative HCT at the time of enrollment
* Female patients who are pregnant are ineligible as many of the medications used in this protocol could be harmful to unborn children and infants
* Sexually active patients of reproductive potential who have not agreed to use an effective contraceptive method for the duration of their study participation
* PATIENT EXCLUSION CRITERIA TO PROCEED TO HCT:
* Patients with uncontrolled fungal, bacterial, viral, or parasitic infections are excluded. Patients with history of fungal disease during chemotherapy may proceed if they have a significant response to antifungal therapy with no or minimal evidence of disease remaining by computed tomography (CT) evaluation
* Patients with active central nervous system (CNS) leukemia or any other active site of extramedullary disease at the time of initiation of the conditioning regimen are not permitted.

  * Note: Those with prior history of CNS or extramedullary disease, but with no active disease at the time of pre-transplant workup, are eligible
* Pregnant or breastfeeding females are ineligible as many of the medications used in this protocol could be harmful to unborn children and infants

Ages: 6 Months to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 435 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Severe GVHD (Grade III-IV acute GVHD or chronic GVHD requiring systemic immunosuppressive therapy) | Up-to 1-year post hematopoietic cell transplantation (HCT)
  We will estimate the cumulative incidence of severe GVHD at 1-year post-HCT and corresponding 95% confidence interval among enrolled and eligible patients randomly assigned to either HAPLO or MUD arms who actually undergo HCT.
Disease free survival (DFS) (where an event is the occurrence of death from any cause or relapse) | From date of randomization to up-to 1 year post randomization
  We will estimate the cumulative incidence at 1 year post randomization and the corresponding 95% confidence interval among all enrolled and eligible patients randomly assigned to either HAPLO or MUD arms.

SECONDARY OUTCOMES:
Overall survival (OS) | From date of randomization to up-to 1-year post-HCT
  We will estimate the cumulative incidence of all-cause mortality events up-to 1-year post-HCT and the corresponding 95% confidence interval among all enrolled, eligible, randomized patients.
Summary score from the Generic Pediatric Quality of Life Inventory (PedsQL) (excluding School Functioning) | At 6-months, 1 year and 2 years post-HCT
  For enrolled, eligible patients who consent to optional QoL studies, we will estimate the mean PedsQL score (excluding School Functioning) among patients randomized to the Haplo arm, the MUD arm, and among patients who enroll to arm C. For each, we will also calculate a corresponding 95% confidence interval.
Summary score from the PedsQL Stem Cell Transplant module | 6-months, 1 year and 2 years post-HCT
  For enrolled, eligible patients who consent to optional QoL studies, we will estimate the mean PedsQL Stem Cell Transplant module score among patients randomized to the Haplo arm and the MUD arm, and among patients who enroll to arm C. For each, we will calculate a corresponding 95% confidence interval.

OTHER OUTCOMES:
Neutrophil engraftment (defined as achieving a donor derived absolute neutrophil count (ANC) >= 500/uL for three consecutive measurements on different days) | Day 30 and Day 100 post-transplant
  We will estimate the cumulative incidences of neutrophil engraftment by Day 30 and Day 100 post-HCT and corresponding 95% confidence intervals among enrolled, eligible patients randomized to either the Haplo or MUD arm and who undergo HCT.
Platelet engraftment (defined as the first day of a minimum of three consecutive measurements on different days such that the patient has achieved a platelet count > 20,000/μL and > 50,000/μL with no platelet transfusions in the preceding seven days) | Day 30 and Day 100 post-transplant
  We will estimate cumulative incidences of platelet engraftment by Day 30 and Day 100 post-HCT and corresponding 95% confidence intervals among enrolled, eligible patients randomized to either the Haplo or MUD arms and who undergo HCT.
Primary and secondary graft failure | 60 days post transplant
  Primary (defined as lack of donor-derived neutrophil engraftment) and secondary graft failure (defined as initial donor-derived neutrophil engraftment followed by subsequent decline in ANC to < 500/μL with loss of donor chimerism to < 10% donor CD3 in peripheral blood or bone marrow). We will estimate cumulative incidences of primary and separately, secondary graft failure by Day 60 post-HCT and corresponding 95% confidence intervals among enrolled, eligible patients randomized to either Haplo or MUD arms and who undergo HCT.
Acute graft versus host disease (aGVHD) Grades II-IV and III-IV | Day 100 and Day 180 post-HCT
  We will estimate cumulative incidences of Grade II-IV aGVHD and separately, Grade III-IV aGVHD by Days 100 and 180 post-HCT and corresponding 95% confidence intervals among enrolled, eligible patients randomized to either Haplo or MUD arms and who undergo HCT.
Transplant related mortality (TRM) | 6-months, 1, and 2-year post-HCT
  We will estimate cumulative incidences of transplant-related mortality by 6-months, 1-year, and 2-years post-HCT and corresponding 95% confidence intervals among enrolled, eligible patients randomized to either Haplo or MUD arms and who undergo HCT.
Relapse | 6-months, 1, and 2-years post-HCT
  We will estimate cumulative incidences of relapse by 6-months, 1-year, and 2-years post-HCT and corresponding 95% confidence intervals among enrolled, eligible patients randomized to either Haplo or MUD arms.
Graft-versus-host disease (GVHD)-free relapse-free survival (GRFS) (using the standard definition and two landmark definitions) | 1-year, 18-months, and 2-years post-HCT
  We will estimate cumulative incidences of GRFS events using all three definitions by 1-year, 18-months, and 2-years post-HCT and corresponding 95% confidence intervals among enrolled, eligible patients randomized to either Haplo or MUD arms and who undergo HCT.
Mild, moderate, and severe chronic graft versus host disease (cGVHD) | 6-months, 1, and 2-year post-HCT
  We will estimate cumulative incidences of mild, moderate, and severe cGvHD by 6-months, 1-year, and 2-years post-HCT and corresponding 95% confidence intervals among enrolled, eligible patients randomized to either Haplo or MUD arms and who undergo HCT.
Significant fungal infections (defined as proven or probable fungal infection according to the De-Pauw definition) | Up-to 1-year post-HCT
  We will estimate the cumulative incidence of significant fungal infections by 1-year post-HCT and the corresponding 95% confidence interval among enrolled, eligible patients randomized to either Haplo or MUD arms.
Viremia (with or without end organ disease) requiring hospitalization and/or systemic antiviral therapy | Up to 1-year post-HCT
  We will estimate the cumulative incidence of viremia by 1-year post-HCT and the corresponding 95% confidence interval among enrolled, eligible patients randomized to either Haplo or MUD arms.
Sinusoidal obstruction syndrome (SOS) (defined by the Cairo criteria and, separately, the EBMT, Baltimore, and modified Seattle criteria) | Up to 100-days post-HCT
  We will estimate the proportion of patients experiencing SOS under the separate definitions by 100-days post-HCT and the corresponding 95% confidence interval among enrolled, eligible patients randomized to either Haplo or MUD arms.
Transplant-associated thrombotic microangiopathy (TA-TMA) | Up to 100-days post-HCT
  We will estimate the proportion of TA-TMA events up-to 100-days post-HCT and the corresponding 95% confidence interval among enrolled, eligible patients randomized to either Haplo or MUD arms and who undergo HCT.
Reconstitution of T, B, and natural killer (NK) cells and immunoglobulins | At 30-days, 60-days, 100-days, 180-days and 365-days after HCT
  We will estimate the median of the distribution of T, B, NK cells, and immunoglobulins among patients given each of three HCT methods (Haplo PTCy, Haplo alpha-beta T-cell depletion, and MUD).
Vaccination-specific antibody titers | 12-18 months post-HSCT
  We will estimate theedian antibody titer among patients given each of three HCT methods (haplo PTCy, haplo alpha-beta T-cell depletion, and MUD).
Resource utilization (defined using the length of HCT hospital stay including readmissions within 100-days post-HCT, and using costs (inpatient) within the first 100-days and 2-years post HCT using Public Health Information System) | 100-days and 2-years post-HCT
  The average proportion of days spent hospitalized will be computed for patients randomized to the Haplo and MUD arms and corresponding 95% confidence intervals will be reported. The median inpatient PHIS adjusted costs by day 100 and 2-years post-HCT will be calculated for patients randomized to Haplo and MUD arms.
incorporating total body irradiation (TBI) delivered with volumetric modulated arc therapy (VMAT) or tomotherapy | Date of initiating TBI through 100 days post-transplant.
  Will be assessed by quality assurance monitoring. Will review treatment plans along with treatment received using data submitted to IROC and will describe the proportion of patients whose planned and actual TBI treatments align among those who received VMAT or tomotherapy. Will quantify the proportion of patients receiving VMAT or tomotherapy TBI who experience serious adverse events (defined as any AE reported through CTEP-AERS) and, separately, who experience any unexpected AE. Will estimate the cumulative incidence of death or relapse (DFS as a composite event) as well as death and relapse separately, and TRM by 0.5, 1, and 2-years year post-transplant from the time of starting TBI among those who receive VMAT or tomotherapy. For relapse and TRM, competing risk analysis will be used, as described under 9.3.5.1. 95% confidence intervals for each of these point estimates will also be provided.

CONTACTS AND LOCATIONS:
Overall Officials: Heather J Symons, Principal Investigator — Children's Oncology Group
Locations (63):
- United States (57):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Norton Children's Hospital, Louisville, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospital of Michigan, Detroit, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
- The Children's Hospital at Westmead, Westmead, New South Wales, Australia
- Canada (5):
  - Alberta Children's Hospital, Calgary, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec